CLINICAL TRIAL: NCT01393041
Title: Clinical Study of the St. Jude Medical Angio-Seal VIP Vascular Closure Device Following Diagnostic and/or Interventional Endovascular Procedures
Brief Title: St. Jude Medical Angio-Seal VIP Vascular Closure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901
Record Dates: First submitted 2011-06-22; First posted 2011-07-13 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Patients Requiring a Diagnostic and/or Interventional Diagnostic Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Angio-Seal VIP (Other)
  Interventions: Device: Angio-Seal VIP

INTERVENTIONS:
Device: Angio-Seal VIP — Vascular Closure Device

SUMMARY:
The purpose of this clinical study is to assess device deployment characteristics and performance, as well as adverse events (vascular complications) of the SJM Angio-Seal VIP 6 French device utilizing the SJM collagen.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing a diagnostic and/or interventional endovascular procedure via a retrograde femoral arterial access.
2. Patient is of legal age.
3. Patient has given written informed consent for participation prior to the procedure.
4. Patient is willing to undergo all study procedures and adhere to data collection and follow-up requirements.

Exclusion Criteria:

1. Patient is unable to provide written informed consent.
2. Patient has an inability or is unwilling to adhere to data collection and follow-up requirements.
3. Patients who are pregnant or lactating.
4. Patient may not participate in another clinical trial which has the potential to impact hemostasis (pharmaceutical/ device/ homeopathic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Device deployment characteristics and performance | At procedure
  Device Deployment Success and rationale for non-deployment, procedural circumstances present during deployment such as type of procedure and procedure duration, Time to hemostasis, and assessment of vascular complications prior to leaving the cath lab. Data will be summarized using descriptive statistics in addition to listings or summary data tables being provided.
Adverse events (vascular complications) | Ongoing
  Adverse events (vascular complications) out to 30 days post-procedure on patients who have undegone a diagnostic and/or interventional procedure.

SECONDARY OUTCOMES:
Time to hemostasis | The time elapsed from device deployment (cutting of the suture) to complete cessation of arterial bleeding, stratified as hemostasis in less than 1 minute, 1-5 minutes, or greater than 5 minutes.
Rate of minor vascular complications | Ongoing

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Luedenscheid, Lüdenscheid, Germany